CLINICAL TRIAL: NCT07212400
Title: Collection of Stool From Healthy Donors for the ex Vivo Study of Shifts of Microbiome Induced by Dairy Phages and Antibiotics: a Model of Bacteria/Host Interaction
Brief Title: Collection of Stool From Healthy Donors for the ex Vivo Study of Shifts of Microbiome Induced by Dairy Phages and Antibiotics: a Model of Bacteria/Host Interaction (DAIRY-SHAPE)
Acronym: DAIRY-SHAPE
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00701-48
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: General Population (no Specific Condition or Disease)
Keywords: phages, antibiotics
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The gut microbiota plays a crucial role in health through its involvement in pathogen defense, immune regulation, and nutrient digestion. Microbiota diversity is essential to maintain these functions, and disturbances caused by antibiotic intake or extreme diets can lead to an imbalance (dysbiosis), which is often described as being implicated in numerous diseases as well as in the proliferation of antibiotic-resistant pathogens.

The microbiota is defined as the community of microorganisms inhabiting the intestine, including bacteria, viruses, and bacteriophages (phages). These phages, through their ability to destroy the bacteria they infect, play an important role in regulating bacterial populations and could therefore be essential for restoring balance and diversity in the gut.

Probiotics, foods that support the microbiota such as dairy products, are of particular interest because the specific interactions between phages and bacteria within these food microbiomes could stimulate microbiota restoration.

This study aims to evaluate the effectiveness of phage-based functional foods in restoring intestinal homeostasis and, by extension, improving human health. It will serve as a model to examine how phages present in foods, particularly dairy products, influence gut microbial diversity and to determine whether these phages promote recovery after antibiotic-induced disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 60 years
* Varied and balanced omnivorous diet

Exclusion Criteria:

* Vegetarian, vegan, or restrictive diet
* Use of medications (antibiotics, anti-inflammatory drugs, immunosuppressants, and/or probiotics, prebiotics, or synbiotics), either as drugs or dietary supplements, within the 3 months prior to sample collection
* Pregnant and/or breastfeeding women
* Presence of an acute or chronic disease (gastrointestinal, metabolic, immune, or inflammatory), diagnosed or suspected
* Colonoscopy within the past 3 months
* Known food allergy or intolerance (e.g., gluten, lactose, FODMAPs) that may alter the usual diet and/or microbiota composition
* Individuals under legal protection (guardianship, trusteeship, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General population residing in Paris Region (Ile-de-France)
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2028-11-16 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | Up to 3 years
  To assess the ability of dairy phages to modulate the intestinal microbiota in vitro using a fermenter system, in the presence and absence of antibiotics.
Secondary Outcome | Up to 3 years
  To monitor the temporal dynamics of the intestinal microbiota following the addition of dairy phages and antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Eugen PFEIFER, Dr., Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Metagenopolis, Jouy-en-Josas, France

IPD SHARING:
Plan to Share IPD: No